CLINICAL TRIAL: NCT01498120
Title: An Open-Label, Long-Term, Follow-Up Study To Determine The Safety, Tolerability, and Efficacy of Rotigotine Transdermal System As Monotherapy in Adolescents With Restless Legs Syndrome
Brief Title: Long-Term Follow-Up Study for Safety, Efficacy and Tolerability of Rotigotine in Adolescents With Restless Legs Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP1005
Record Dates: First submitted 2011-12-16; First posted 2011-12-23 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Restless Legs Syndrome
Keywords: Rotigotine; Restless Legs Syndrome; RLS; Long-term; Adolescents
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rotigotine (Experimental): Optimal dose after titration period
  0.5 mg/24 h (2.5 cm^2)- 1 mg/24 h (5 cm^2)- 2 mg/24 h (10 cm^2)- 3 mg/24 h (15 cm^2)
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Optimal dose after titration period
  0.5 mg/24 h (2.5 cm^2)- 1 mg/24 h (5 cm^2)- 2 mg/24 h (10 cm^2)- 3 mg/24 h (15 cm^2)
  1 patch /day

SUMMARY:
This is a Phase 2, multicenter, open-label, single-arm, optimal dose, long-term follow-up study of monotherapy administration of rotigotine transdermal patch in adolescents with Restless Legs Syndrome (RLS). This study will assess the long-term safety and tolerability of Rotigotine treatment in adolescents with RLS.

DETAILED DESCRIPTION:
Study design was changed and an amendment was prepared accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Tolerated the first dose level of Rotigotine in a previous study in adolescents with Restless Legs Syndrome (RLS), without meeting withdrawal criteria
* Is expected to benefit from participation, in the opinion of the investigator
* Subject/legal representative is considered reliable and capable of adhering to the protocol, visit schedule, and study patch application/removal, according to the judgment of the investigator

Exclusion Criteria:

* Previously participated in this study
* Is experiencing an ongoing serious adverse event (SAE) that is assessed to be related to Rotigotine by the investigator or sponsor
* Pregnant or nursing or is a female of childbearing potential who is not surgically sterile or does not consistently use 2 combined medically acceptable methods of birth control (including at least 1 barrier method), unless not sexually active
* Any medical or psychiatric condition that, in the opinion of the investigator, can jeopardize or would compromise the subject's ability to participate
* Active suicidal ideation as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Since the Last Visit" version of the Columbia Suicide Severity Rating Scale (C-SSRS) of the final evaluation visit of the previous Rotigotine study

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 1-877-822-9493 (UCB)
Locations (5):
- United States (5):
  - 012, Los Angeles, California
  - 009, Orange, California
  - 014, Spring Hill, Florida
  - 013, Indianapolis, Indiana
  - 001, Destrehan, Louisiana

REFERENCES:
- See also: Product Information — https://www.neupro.com/neupro-prescribing-information.pdf?v=1489766618
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in USA in January 2012 and concluded in December 2015.
Pre-assignment Details: Participant Flow refers to the Safety Set (SS) which consists of all subjects who were randomized in this study and received at least 1 dose of study medication.
Groups:
- Rotigotine: Adolescent subjects who were previously administered rotigotine transdermal system (Neupro) in study SP1004 (NCT01495793), received the rotigotine transdermal patch in the following doses and sizes: 0.5mg/24h (2.5cm^2), 1mg/24h (5cm^2), 2mg/24h (10cm^2) and 3mg/24h (15cm^2).
Period: Overall Study
Arm/Group | Rotigotine
Started | 14
Completed | 1
Not Completed | 13
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 5
Not completed — AE, non-serious non-fatal | 3
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: All enrolled subjects who received at least 1 dose of study medication were included in the SS.
Arm/Group | Rotigotine
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.4 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Withdrawn Due to An Adverse Event (AE) From Visit 1 (Day 1) Through End of Study
Description: An Adverse Event is any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: Visit 1 (Day 1) through End of Study (approximately 2 years)
Population: All enrolled subjects who received at least 1 dose of study medication were included in the SS.
Measure: Number; unit: subjects
Groups:
- Rotigotine (Safety Set): The Safety Set (SS) which consists of all subjects who were randomized in this study and received at least 1 dose of study medication. Adolescent subjects who were previously administered rotigotine transdermal system (Neupro) in study SP1004 (NCT01495793), received the rotigotine transdermal patch in the following doses and sizes: 0.5mg/24h (2.5cm^2), 1mg/24h (5cm^2), 2mg/24h (10cm^2) and 3mg/24h (15cm^2).
Arm/Group | Rotigotine (Safety Set)
Number analyzed (Participants) | 14
subjects | 3

2. Primary Outcome: Number of Subjects With At Least One Adverse Event (AE) From Visit 1 (Day 1) to End of Study
Description: as for outcome 1
Time Frame: From Visit 1 (Day 1) through End of Study (approximately 2 years)
Population: All enrolled subjects who received at least 1 dose of study medication were included in the SS.
Measure: Number; unit: subjects
Arm/Group | Rotigotine (Safety Set)
Number analyzed (Participants) | 14
subjects | 10

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Visit 1 (Week 0) until Safety Follow Up Visit (up to 25 months).
Description: All enrolled subjects who received at least 1 dose of study medication were included in the SS.
Arm/Group | Rotigotine (Safety Set)
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 10/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (Safety Set) (N=14)
Palpitations (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (7)
Vomiting (Gastrointestinal disorders) | 3 (6)
Application site pruritus (General disorders) | 1 (1)
Febrile disorders (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Blood sodium increased (Investigations) | 1 (1)
Toxicology laboratory analyses (Investigations) | 1 (1)
Drug screen positive (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (3)
Dizziness (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Sudden onset of sleep (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Enuresis (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days